CLINICAL TRIAL: NCT04644224
Title: A Peer and Family-Based Approach to Obesity in African American Families
Brief Title: Parent and Family Oriented Support Interventions for the Facilitation of Weight Loss in African American Families
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2017-0827; NCI-2020-07645 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2017-0827 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2020-10-21; First posted 2020-11-25 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Obesity-Related Malignant Neoplasm
MeSH Terms: interventions — Early Intervention, Educational; Educational Status; Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group I (coaching session, navigation session, support group) (Experimental): Parents/caregivers whose churches are randomized to Group I, attend monthly health coaching sessions over 1 hour each for 12 months, 9 resource navigation sessions over 12 months, and monthly support groups for 12 months.
  Interventions: Other: Educational Activity; Other: Educational Intervention; Other: Questionnaire Administration; Procedure: Support Group Therapy
- Group II (coaching session, navigation session, support group) (Experimental): Families whose churches are randomized to Group II, attend monthly health coaching sessions over 1 hour each for 12 months, 9 resource navigation sessions over 12 months, and monthly support groups for 12 months.
  Interventions: Other: Educational Activity; Other: Educational Intervention; Other: Questionnaire Administration; Procedure: Support Group Therapy
- Group III (educational handbook) (Active Comparator): Families whose churches are randomized to Group III, receive an educational handbook on cancer prevention.
  Interventions: Other: Informational Intervention; Other: Questionnaire Administration

INTERVENTIONS:
Other: Educational Activity — Attend health coaching session
  Arms: Group I (coaching session, navigation session, support group); Group II (coaching session, navigation session, support group)
Other: Educational Intervention — Attend resource navigation session
  Other Names: Education for Intervention; Intervention by Education; Intervention through Education; Intervention, Educational
  Arms: Group I (coaching session, navigation session, support group); Group II (coaching session, navigation session, support group)
Other: Informational Intervention — Receive handbook
  Arms: Group III (educational handbook)
Other: Questionnaire Administration — Ancillary studies
Procedure: Support Group Therapy — Attend support group
  Arms: Group I (coaching session, navigation session, support group); Group II (coaching session, navigation session, support group)

SUMMARY:
This study tests the effectiveness of parent and family oriented support interventions that are designed to help with weight loss among African American families. Obesity tends to run in families, thus family based interventions, with parents as main change agents have been strongly recommended. The parent and family oriented support Interventions may help facilitate weight loss among African American families.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine whether a parent/caregiver intervention or a family intervention can produce greater weight loss among obese African American (AA) parents at 12 months compared to a cancer prevention group (control).

II. Use the Reach, Effectiveness, Adoption, Implementation, and Maintenance (RE-AIM) model, to evaluate individual and church-level barriers and facilitators on program reach, effectiveness, adoption, implementation, maintenance and dissemination.

SECONDARY OBJECTIVES:

I. Explore whether a parent/caregiver intervention and a family intervention can produce weight maintenance or weight loss, as determined by change in body mass index (BMI) z-score, among AA children at risk for obesity at 12 months compared to the control group.

II. Determine the extent to which the proposed interventions improve fruit and vegetable (FV) consumption, physical activity, blood pressure, body fat percentage, muscle mass and waist circumference.

OUTLINE: Churches are randomized to 1 of 3 groups.

GROUP I: Parents/caregivers whose churches are randomized to Group I, attend monthly health coaching sessions over 1 hour each for 12 months, 9 resource navigation sessions over 12 months, and monthly support groups for 12 months.

GROUP II: Families whose churches are randomized to Group II, attend monthly health coaching sessions over 1 hour each for 12 months, 9 resource navigation sessions over 12 months, and monthly support groups for 12 months.

GROUP III: Families whose churches are randomized to Group III, receive an educational handbook on cancer prevention.

ELIGIBILITY:
Inclusion Criteria:

* DYAD: Be parent/caregiver (legal parent or custodial grandparent; male or female) and child willing to participate
* DYAD: Live together in the same household
* PARENT/CAREGIVER: Self-identify as a racial ethic minority (i.e., black or African American or Hispanic)
* PARENT/CAREGIVER: Parent or caregiver age 18 through 65 years old
* PARENT/CAREGIVER: Are overweight (BMI greater than or equal to 25);
* PARENT/CAREGIVER: Are not currently participating in a physical activity (PA), diet, or weight management program
* PARENT/CAREGIVER: Have a valid home address, telephone number, and internet access
* PARENT/CAREGIVER: Enroll with a child aged 8-17 years
* PARENT/CAREGIVER: Are able to speak English

Exclusion Criteria:

* PARENT/CAREGIVER: They are currently pregnant or thinking about becoming pregnant during the study period
* PARENT/CAREGIVER: They present any contraindications for exercise based on responses to the PA Readiness Questionnaire plus (PAR-Q +)

Exclusion criteria for child:

1) None.

Ages: 10 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2019-01-17 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Weight loss of parents | Up to 18 months
  Will use the generalized linear mixed model (GLMM) regression, which takes into account both within-cluster (e.g., within church) and, as applicable, within-individual (e.g., overtime) correlations between observations of each primary and secondary outcomes of interest.
Reach (Part 1 of the RE-AIM framework) | Up to 18 months
  Measured as the number of churches invited to participate, number enrolled, and differences between the two groups.
Effectiveness (Part 2 of the RE-AIM framework) | Up to 18 months
  Measured as the impact on weight loss: 6 focus groups and 15 individual interviews at 18 months to understand unanticipated outcomes; interview lay health workers (LHWs) about implementation.
Adoption (Part 3 of the RE-AIM framework) | Up to 18 months
  Will be measured by asking churches about factors that helped or hindered adoption or implementation and will they adopt intervention when completed.
Implementation (Part 4 of the RE-AIM framework) | Up to 18 months
  Measured as study attendance and assessments, number of health coaching, LHW and support group sessions, number of staff training, and self-monitoring practices.
Maintenance (Part 5 of the RE-AIM framework) | Up to 18 months
  Long-term maintenance in parent/families at 18 months measured by family and church attrition, to assess church's ability to maintain employment of LHWs and their willingness to remain in this role.

SECONDARY OUTCOMES:
Child's body mass index (BMI) z-score | Up to 18 months
  Will use the GLMM regression, which takes into account both within-cluster (e.g., within church) and, as applicable, within-individual (e.g., overtime) correlations between observations of each primary and secondary outcomes of interest.
Fruit and vegetable consumption | Up to 18 months
  Will use the GLMM regression, which takes into account both within-cluster (e.g., within church) and, as applicable, within-individual (e.g., overtime) correlations between observations of each primary and secondary outcomes of interest.
Physical activity | Up to 18 months
  Will use the GLMM regression, which takes into account both within-cluster (e.g., within church) and, as applicable, within-individual (e.g., overtime) correlations between observations of each primary and secondary outcomes of interest.
Blood pressure | Up to 18 months
  Will use the GLMM regression, which takes into account both within-cluster (e.g., within church) and, as applicable, within-individual (e.g., overtime) correlations between observations of each primary and secondary outcomes of interest.
Body fat percentage | Up to 18 months
  Will use the GLMM regression, which takes into account both within-cluster (e.g., within church) and, as applicable, within-individual (e.g., overtime) correlations between observations of each primary and secondary outcomes of interest.
Waist circumference | Up to 18 months
  Will use the GLMM regression, which takes into account both within-cluster (e.g., within church) and, as applicable, within-individual (e.g., overtime) correlations between observations of each primary and secondary outcomes of interest.

CONTACTS AND LOCATIONS:
Overall Officials: Lorna McNeill, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org

DOCUMENTS (1):
  • Informed Consent Form (2025-03-24): https://cdn.clinicaltrials.gov/large-docs/24/NCT04644224/ICF_000.pdf